CLINICAL TRIAL: NCT02166515
Title: The Study of Massively Parallel Sequencing in Early Detection for Gynecologic Malignant Tumor
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zhiqing, Liang (Other)
Collaborators: Shenzhen Huada Genomics Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Zhiqing, Liang, Department of Obstetrics and Gynaecology, Southwest Hospital, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: 001; fck001 (Registry Identifier: ZLiang)
Record Dates: First submitted 2014-02-10; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Gynecologic Malignant Tumor
Keywords: cervical cancer; ovarian cancer; endometrial cancer; high-throughput sequencing
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The sample of blood, urine, cervical exfoliated cells and cancer tissue of patient should be used only in this research with informed consent. The remaining part will be Safekeeping.All information is strictly confidential.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- experiment group: patients with cervical cancer, endometrial cancers or ovary cancer
- control group: postmenopausal women with benign tumor

SUMMARY:
As human aging, 50% of women will be faced with the threat of cancer, especially gynecological malignancies. Ovarian, cervical and endometrial cancer are three major gynecological malignancies. In recent years, the incidence of cervical cancer, especially in young women significantly increased; ovarian cancer, although the incidence of malignant tumors in the female reproductive system ranked second, but its mortality rate already in the first place; and the morbidity and mortality of endometrial cancer is also rising.

The key to gynecologic malignancies is how to early diagnose and treat. With the advancement of science and technology, such as molecular biology techniques widely used in the medical field, early diagnosis, proper treatment and other aspects in gynecologic malignancies is expected to achieve a breakthrough. Genome-wide scan strategy, making the whole genome for linkage analysis for gynecological malignancies possible. Therefore, the investigators intend to find specific mutations to provide a new early screening approach for gynecological malignancies, which in later result in early diagnosis and specific treatment for gynecological malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Female aging from 16 to 75-year old;
* Preoperative diagnosis of gynecologic malignancies;
* Have the ability to comply with Research programs;
* Voluntarily participate in the study and signed an informed consent form

Exclusion Criteria:

* The cases do not meet the inclusion criteria should be removed from,indicating the reason for excluding.

Ages: 16 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The experiment group are patients with cervical cancer, ovarian cancer or endometrial cancer.While the control group are volunteers on the basis of informed consent.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Gene mutation from species of cervical cancer, endometrial cancers and ovary cancer | 4 years
  We expect to found spcific DNA mutation in the species (peripheral blood, liquid Pap smear and cancer tissue) from cervical cancer, endometrial cancers and ovary.

SECONDARY OUTCOMES:
the difference between detection sensitivity | 4 years
  Comparing sensiitivity of the three kinds of samples on early detection of gynecologic malignancies

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Southwest Hospital, Third Military, Chongqing, Chongqing Municipality, China